CLINICAL TRIAL: NCT02643030
Title: The Effect of Hypercapnia on Regional Cerebral Oxygen Saturation in the Sitting Position
Brief Title: Hypercapnia During Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GIRBA2674-2012
Record Dates: First submitted 2015-12-23; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normocapnia (Experimental): Tidal volume (10 ml/kg) and respiratory rate is adjusted to achieve the objective values of ETCO2 35mmHg
  Interventions: Behavioral: normocapnia
- hypercapnia (Active Comparator): Tidal volume (6ml/kg) and respiratory rate is adjusted to achieve the objective values of ETCO2 45mmHg
  Interventions: Behavioral: hypercapnia

INTERVENTIONS:
Behavioral: hypercapnia — Tidal volume (6 ml/kg) and respiratory rate is adjusted to achieve the objective values of ETCO2 45mmHg
  Other Names: ETCO2-45
  Arms: hypercapnia
Behavioral: normocapnia — Tidal volume (10 ml/kg) and respiratory rate is adjusted to achieve the objective values of ETCO2 35mmHg
  Other Names: ETCO2-35
  Arms: normocapnia

SUMMARY:
The purpose of this study is to evaluate the effects of hypercapnia on hemodynamics and cerebral oxygenation during shoulder arthroscopy.

DETAILED DESCRIPTION:
The patients are randomly allocated to receive normocapnia or hypercapnia . After the 70º sitting position, record the mean arterial pressure (MAP), heart rate, and regional oxygen saturation (rSO2).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective shoulder arthroscopic surgery

Exclusion Criteria:

* a history of age > 65 years, morbidly obesity (BMI > 30 kg/m2), diffuse lung disease, uncontrolled systemic hypertension, intracranial disease, cardiovascular and cerebrovascular disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Regional cerebral oxygen saturation | Change from Regional cerebral oxygen saturation at 2,4,6,8,10,20 min after anesthetic induction and sitting position

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, MD, Study Chair — Gachon University Gil Medical Center

REFERENCES:
- [Result] Pohl A, Cullen DJ. Cerebral ischemia during shoulder surgery in the upright position: a case series. J Clin Anesth. 2005 Sep;17(6):463-9. doi: 10.1016/j.jclinane.2004.09.012. PMID 16171668